CLINICAL TRIAL: NCT03162692
Title: Preoperative Anxiety's Incidence and Related Factors in Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Chief physician and Associate Professor, Xuzhou Medical University
Other Study IDs: XYFY2017-KL021-01
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Elective Surgery; Intravenous Anesthesia; Preoperative Anxiety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative anxiety is often described as an uncomfortable, tense unpleasant mood before surgery, an emotional response to a potential challenge or threat to reality. Data show that adult patients with preoperative anxiety rate of 30-40%. The main reason for the occurrence of patients for surgery, anesthesia and other factors of fear. Preoperative anxiety itself is not a mental illness, but studies have confirmed that the occurrence of preoperative anxiety and postoperative complications were positively correlated, and the existence of preoperative anxiety in patients with conventional postoperative analgesic effect is poor. At present, there are still few studies on the relationship between preoperative anxiety and postoperative complications and analgesia. At the same time, there is a lack of large sample size to study the incidence of preoperative anxiety and its related predictors.

DETAILED DESCRIPTION:
Surgical patients often have varying degrees of preoperative anxiety.The aim of this study was to determine the incidence of preoperative anxiety and related predictors, and to evaluate the effect of anxiety on anesthesia and postoperative pain and prognosis. The study also showed that prostaglandin, catecholamines, cortex Effects of alcohol and inflammatory cell level on postoperative pain in patients with preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Sign that informed consent is willing to participate in the study
* Education: primary school and above
* 1 days after elective general anesthesia surgery
* ASA score grade I-III

Exclusion Criteria:

* Emergency surgery
* Severe mental illness patients (such as anxiety, depression, schizophrenia, etc.)
* Taking anti-anxiety or antidepressants (benzodiazepines, tricyclic antidepressants, selective serotonin inhibitors, monoamine oxidase inhibitors, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2000 patients undergoing elective general anesthesia in surgery in Xuzhou Medical University patients.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | All patients are evaluated one day before surgery
  as measured by STAI (state-trait anxiety questionnaire)

SECONDARY OUTCOMES:
VAS pain score | at 3 hours, 6 hours, 24 hours, 48 hours after surgery
  as measured by visual smileys scale

OTHER OUTCOMES:
blood inflammation index | Extraction of arterial blood before anesthesia induction
  extraction of patients with arterial blood to laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Jindong Liu, M.S, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lieb K, Fiebich BL, Berger M. [Substance P receptor antagonists--a new antidepressive and anxiolytic mechanism?]. Nervenarzt. 2000 Sep;71(9):758-61. doi: 10.1007/s001150050661. German. PMID 11042872
- [Result] Maki Y. [A behavioral and neurochemical study on the mechanism of the anxiolytic effect of monoamine oxidase inhibitors]. Hokkaido Igaku Zasshi. 2001 May;76(3):133-42. Japanese. PMID 11481866
- [Result] Yamauchi M, Hiraoka S, Imanishi T. [Role of the serotonergic nervous system in anxiety disorders and the anxiolytic mechanism of selective serotonin reuptake inhibitors]. Nihon Shinkei Seishin Yakurigaku Zasshi. 2006 Nov;26(5-6):193-8. Japanese. PMID 17240844
- [Result] Matsumoto K, Puia G, Dong E, Pinna G. GABA(A) receptor neurotransmission dysfunction in a mouse model of social isolation-induced stress: possible insights into a non-serotonergic mechanism of action of SSRIs in mood and anxiety disorders. Stress. 2007 Mar;10(1):3-12. doi: 10.1080/10253890701200997. PMID 17454962
- [Result] Herrera-Ruiz M, Gonzalez-Carranza A, Zamilpa A, Jimenez-Ferrer E, Huerta-Reyes M, Navarro-Garcia VM. The standardized extract of Loeselia mexicana possesses anxiolytic activity through the gamma-amino butyric acid mechanism. J Ethnopharmacol. 2011 Nov 18;138(2):261-7. doi: 10.1016/j.jep.2011.09.010. Epub 2011 Sep 16. PMID 21979412
- [Result] Mico JA, Prieto R. Elucidating the mechanism of action of pregabalin: alpha(2)delta as a therapeutic target in anxiety. CNS Drugs. 2012 Aug 1;26(8):637-48. doi: 10.2165/11634510-000000000-00000. PMID 22784017
- [Result] O'Donovan A, Slavich GM, Epel ES, Neylan TC. Exaggerated neurobiological sensitivity to threat as a mechanism linking anxiety with increased risk for diseases of aging. Neurosci Biobehav Rev. 2013 Jan;37(1):96-108. doi: 10.1016/j.neubiorev.2012.10.013. Epub 2012 Nov 2. PMID 23127296
- [Result] Fan JM, Chen XQ, Du JZ. Prenatal stress, anxiety and depression: a mechanism involving CRH peptide family. Neuro Endocrinol Lett. 2014;35(6):429-39. PMID 25433848
- [Result] He W, Zhou Q, Yu S, Cai D, Wang Q, Zhang X, Huang WQ. [Mechanism on atrial natriuretic peptide receptor in anti-anxiety with acupuncture based on its tranquilizing effect]. Zhongguo Zhen Jiu. 2015 Jan;35(1):101-4. Chinese. PMID 25906584